CLINICAL TRIAL: NCT01363973
Title: Pilot Study to Evaluate the Efficacy and Safety of Transcutaneous Electrical Stimulation on Swallowing in Patients With Oropharyngeal Dysphagia After Stroke
Brief Title: Effect of Transcutaneous Electrical Stimulation on Post-stroke Dysphagic Patients
Acronym: EETI-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Pere Clave, MD, PhD, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EETI-01
Record Dates: First submitted 2011-05-27; First posted 2011-06-02 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Dysphagia
Keywords: oropharyngeal dysphagia; post-stroke
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sensory stimulation (Experimental): Transcutaneous electrical stimulation at 75% of motor threshold
  Interventions: Device: VITALSTIM transcutaneous electrical stimulation
- Motor stimulation (Experimental): Transcutaneous electrical stimulation at motor threshold
  Interventions: Device: VITALSTIM transcutaneous electrical stimulation

INTERVENTIONS:
Device: VITALSTIM transcutaneous electrical stimulation

SUMMARY:
Oropharyngeal dysphagia (OD, swallowing dysfunction) is a major complaint following stroke. Despite its enormous impact on functional capacity, quality of life, and survival, OD is both underestimated and underdiagnosed as a cause of major nutritional and respiratory complications in stroke patients. A recent systematic review on the effects of rehabilitation therapy on OD concluded that although some positive effects were found, the number of studies was small, many of them had methodological problems and there was a need for further research using randomized controlled trials. Transcutaneous electrical stimulation was approved by the FDA as a treatment of dysphagia in June 2001 and is traditionally used to activate pharyngeal muscles through stimulation of peripheral motor nerves (neuromuscular electrical estimulation, NMES). However, their real effectiveness and safety in the treatment of dysphagia is still matter of discussion (Logemann Dysphagia 2007, Ludlow dysphagia 2007) and studies evaluating NMES therapy, present discordant results. On the other hand, in recent years, transcutaneous electrical stimulation is beginning to use as a sensory strategy (Gallas 2010), avoiding muscle contraction during the treatment.Our research strategy includes the assessment of the therapeutic effect of these two main strategies using transcutaneous electrical stimulation on swallow physiology and clinical outcomes of post-stroke dysphagic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Background of swallowing difficulties associated with stroke, more than 3 months of evolution
* Study explained and signed informed consent

Exclusion Criteria:

* Patients who are suspected or can not meet the protocol. patients who are participating or have participated in a trial last 4 weeks. Patients with active cancer Patients with active infectious process. patients with severe dementia or inability to communicate. patients with neurodegenerative diseases. patients with pacemakers. patients with implanted electrodes. patients with epilepsy or seizure disorders. patients with gastroesophageal reflux.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety of swallow | 5 days
  Prevalence of penetrations or aspirations after the treatment

SECONDARY OUTCOMES:
Efficacy of swallow | 5 days
  Prevalence of residue after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain